CLINICAL TRIAL: NCT07089862
Title: Indobufen Versus Aspirin in Endovascular Unruptured Intracranial Aneurysms Treatment
Brief Title: INdobufen Versus asPirin in Endovascular Unruptured Intracranial Aneurysms Treatment (INPUT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: RenJi Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Jiangnan University Central Hospital (Unknown); Beijing Chao Yang Hospital (Other); Beijing Friendship Hospital (Other); Beijing Shuyi Hospital (Other); The Central Hospital of Lishui City (Other)
Responsible Party: Principal Investigator, Wang Shuo, Director of Department of Cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HX-B-2023016
Record Dates: First submitted 2025-07-22; First posted 2025-07-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Unruptured Intracranial Aneurysm; Indobufen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indobufen+clopidogrel group (Experimental): Patients in the experimental group will be required to take indobufen (100 mg twice daily) + clopidogrel (75 mg once daily) starting 5 days before the procedure and continuing until 180 days postoperatively.
  Interventions: Drug: Indobufen treatment
- Aspirin+clopidogrel group (Active Comparator): Patients in the control group will be required to take aspirin (100 mg once daily) + clopidogrel (75 mg once daily) starting 5 days before the procedure and continuing until 180 days postoperatively.
  Interventions: Drug: Aspirin treatment

INTERVENTIONS:
Drug: Indobufen treatment — Patients in the experimental group will be required to take indobufen (100 mg twice daily) + clopidogrel (75 mg once daily) starting 5 days before the procedure and continuing until 180 days postoperatively.
  Arms: Indobufen+clopidogrel group
Drug: Aspirin treatment — Patients in the control group will be required to take aspirin (100 mg once daily) + clopidogrel (75 mg once daily) starting 5 days before the procedure and continuing until 180 days postoperatively.
  Arms: Aspirin+clopidogrel group

SUMMARY:
This project aims to evaluate the safety and efficacy of the antiplatelet regimen combining indobufen and clopidogrel in preventing ischemic events after stent-assisted coiling embolization and flow diverter implantation for intracranial aneurysms.

Using a randomization system, patients with unruptured intracranial aneurysms scheduled for interventional treatment will be divided into an experimental group and a control group. Patients in the experimental group will be required to take indobufen (100 mg twice daily) + clopidogrel (75 mg once daily) starting 5 days before the procedure and continuing until 180 days postoperatively. Patients in the control group will be required to take aspirin (100 mg once daily) + clopidogrel (75 mg once daily) starting 5 days before the procedure and continuing until 180 days postoperatively.

An independent group of researchers will assess cerebrovascular thromboembolic events and bleeding events at different time points.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years (male or female);
2. Radiologically confirmed saccular intracranial aneurysm (by specialist assessment);
3. Scheduled for endovascular embolization (including: coil embolization with stent assistance or flow diversion);
4. Signed informed consent obtained.

Exclusion Criteria:

1. Concomitant vascular malformations, tumors, abscesses or other cerebral diseases such as multiple sclerosis;
2. Major surgery within 30 days prior to enrollment including fracture surgery or hip replacement;
3. History of ischemic stroke, ischemic heart disease or hemorrhagic disorders including intracranial hemorrhage, gastrointestinal bleeding, fundus hemorrhage or unexplained bleeding within the past 6 months;
4. Planned elective surgery within 3 months after the procedure;
5. Any hematologic disorders or inherited coagulation abnormalities;
6. Severe renal or hepatic dysfunction;
7. History of hemostatic disorders, systemic bleeding, thrombocytopenia or neutropenia;
8. History of symptomatic non-traumatic intracranial hemorrhage or cerebral amyloid angiopathy;
9. Severe cardiopulmonary diseases considered by investigators to be unsuitable for the study;
10. Women of childbearing potential with negative pregnancy test but refusing contraceptive measures, or those who are pregnant or lactating;
11. Current participation in other investigational drug or device trials.

Withdrawal Criteria:

1. Receiving aneurysm treatment other than coil embolization with stent assistance or flow diversion;
2. Occurrence of endpoint events during stent-assisted aneurysm embolization procedure (as adjudicated by the Clinical Events Committee), including procedure-related hemorrhagic events (aneurysm rupture, parent artery rupture, subarachnoid hemorrhage, acute ipsilateral intracerebral hemorrhage, and acute ipsilateral subdural/epidural hematoma) or ischemic events (acute large vessel occlusion, in-stent thrombosis, and diffuse ipsilateral vascular infarction caused by plaque dislodgement);
3. Device-related quality issues during stent-assisted embolization, including stent problems (stent fracture, failure to deploy properly, incomplete expansion due to product defect) and coil problems (premature detachment before intentional deployment, coil unraveling, and failure to detach);
4. Postoperative life expectancy <3 months;
5. Inability to complete 5-day premedication due to emergency surgery or other reasons;
6. Intolerance to oral antiplatelet therapy due to allergy or other contraindications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint Events: Cerebrovascular thromboembolic events occurring within 90 days postoperatively | within 90 days after endovascular treatment of unruptured intracranial aneurysms
  Cerebrovascular thromboembolic events within 90 days after endovascular treatment of unruptured intracranial aneurysms, including: Ischemic stroke, Transient ischemic attack (TIA), Stent thrombosis, Emergency revascularization, Cerebrovascular death
Primary Safety Endpoint Events: Incidence of bleeding events classified as Type 2, 3, or 5 according to the Bleeding Academic Research Consortium (BARC) criteria within 90 days after endovascular treatment of unruptured intracranial aneurysms. | Within 90 days after endovascular treatment of unruptured intracranial aneurysms.
  Bleeding events classified as Type 2, 3, or 5 according to the Bleeding Academic Research Consortium (BARC) criteria within 90 days after endovascular treatment of unruptured intracranial aneurysms.

SECONDARY OUTCOMES:
Cerebrovascular thromboembolic events occurring within 30 days postoperatively | Within 30 days postoperatively
  Cerebrovascular thromboembolic events within 30 days after endovascular treatment of unruptured intracranial aneurysms, including: Ischemic stroke, Transient ischemic attack (TIA), Stent thrombosis, Emergency revascularization, Cerebrovascular death
Cerebrovascular thromboembolic events occurring within 180 days postoperatively | Within 180 days postoperatively
  Cerebrovascular thromboembolic events within 180 days after endovascular treatment of unruptured intracranial aneurysms, including: Ischemic stroke, Transient ischemic attack (TIA), Stent thrombosis, Emergency revascularization, Cerebrovascular death
Platelet aggregation rate within 24 hours before surgery | Within 24 hours before surgery
  Platelet aggregation rate within 24 hours before surgery, including ADP-induced platelet aggregation, Collagen-induced platelet aggregation and Arachidonic acid-induced platelet aggregation.